CLINICAL TRIAL: NCT07205237
Title: Effect of Eliminating Red Meat Consumption on the Cardiovascular System - A Longitudinal Study
Brief Title: Effect of Eliminating Red Meat Consumption on the Cardiovascular System
Acronym: ERRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Clara Rocha (Other)
Responsible Party: Sponsor-Investigator, Maria Clara Rocha, Professor, Escola Superior de Tecnologia da Saúde de Coimbra
Organization: Escola Superior de Tecnologia da Saúde de Coimbra (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ERRM2025
Record Dates: First submitted 2025-07-21; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular (CV) Risk
Keywords: Red meat; Processed meat; Omnivorous; Carotid disease; Lipid changes
MeSH Terms: interventions — Diet; Dyrk Kinases

STUDY DESIGN:
Intervention Model Description: A single-group longitudinal study design was adopted, comprising a 4-week intervention period. Each participant was submitted to 2 evaluation times: at baseline (T0), 4 weeks after eliminating red/processed meat from the diet (T1). The sample was obtained into two different laboratories, in each of which different parameters were assessed: Haematological and Vascular parameters.
  After clarification of the study and signed informed consent, participants were asked to complete a questionnaire containing information on sociodemographic parameters (gender, age, weight and height), behavioural parameters (diet, smoking, alcohol consumption, coffee, vitamin B12 supplements and energy drinks consumption and sports practice) and clinical parameters (use of oral contraception, medication, anaemia, hypertension, cholesterol, diabetes and personal history of CVD). Participants were also instructed to replace red and processed meat from their daily diet, replacing it with fish, eggs or white meat.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group - Diet without Red and Processed Meat (Experimental): All participants follow a four-week diet excluding red and processed meat. Vascular, biochemical, and hematological parameters are assessed at baseline and post-intervention.
  Interventions: Dietary Supplement: Diet without Red and Processed Meat

INTERVENTIONS:
Dietary Supplement: Diet without Red and Processed Meat — Participants replaced red and processed meat in their daily diet with fish, eggs, or white meat, while keeping the food proportions of their meals unchanged.

SUMMARY:
The objective of this clinical trial is to evaluate, in clinically healthy young omnivores, whether excluding red and processed meat from their diets for four weeks results in:

* measurable changes in arterial structure and function;
* measurable changes in key metabolic parameters.

The sample consisted of clinically healthy young people who had been following an omnivorous diet for at least one year. Those with a history that could influence the results were excluded. Exclusion criteria included alcohol or coffee abuse, vitamin B12 supplement intake, anemia, hypertension, cholesterol, diabetes, a history of cardiovascular disease, or an unstable clinical situation. Participants taking chronic medication, except those using oral contraceptives, were also excluded.

A single-group longitudinal study design is adopted, comprising a 4-week intervention period. Each participant undergoes two assessments: at baseline (T0) and 4 weeks after eliminating red/processed meat from the diet (T1). After being informed about the study and signing the informed consent form, participants are asked to complete a questionnaire containing information on sociodemographic (sex, age, weight, and height), behavioral (diet, smoking, alcohol consumption, coffee, vitamin B12 supplements, energy drinks, and sports activity), and clinical parameters (use of oral contraceptives, medications, anemia, hypertension, cholesterol, diabetes, and personal history of CVD). Participants are also instructed to replace red and processed meat in their daily diet with fish, eggs, or white meat, and to maintain the food proportions of their meals unchanged.

DETAILED DESCRIPTION:
Biochemical and Haematological parameters:

To determine blood parameters, 10 ml of peripheral blood was collected by venipuncture for serum and plasma in K3EDTA tubes. The biochemical profile was determined spectrophotometrically on a Prestige 24i chemistry analyzer (Tokyo Boeky, Tokyo, Japan) with reagents from Cormay® (Warsaw, Poland). Complete blood counts are performed on a Cell-Dyn Sapphire™ hematology analyzer (Abbott Laboratories, Santa Clara, CA, USA).

Approximately 7 mL of venous blood is collected per sample in a dry gel tube and centrifuged under vacuum at 1800 g, 4°C for 10 minutes. The serum is then separated into aliquots and stored at -20°C until the desired parameters are achieved. The analytical parameters total cholesterol, HDL-C, LDL-C, triglycerides, and glucose are obtained using the corresponding kit from Cormay, Poland. Concentrations are assessed spectrophotometrically according to the protocol and using the Prestige 24i equipment (TOKYO BOEKI MEDICAL SYSTEM LTD, Tokyo, Japan). The K3EDTA tube is used to perform complete blood counts on the Cell-Dyn Sapphire™ equipment (Abbott Laboratories, Santa Clara, CA, USA). All tests were validated and subjected to quality control.

Vascular parameters:

Participants are placed in the supine position and have a 5-minute rest period before data collection. Subsequently, heart rate (HR), systolic blood pressure (SBP), and diastolic blood pressure (DBP) are measured. The cuff is placed on the right arm, aligned with the brachial artery, and adjusted to the arm circumference.

The common carotid artery (CCA) is assessed using a GE® Vivid T8 ultrasound device with a 6-12 MHz linear probe. The participant is placed in the supine position with the neck in slight hyperextension. A longitudinal section of the CCA is taken, and the image is saved for measurement of systolic (SD) and diastolic diameters (DD) and intima-media thickness (IMT). Subsequently, peak systolic (PSV) and endodiastolic (ED) velocities of the CCA are recorded using pulsed Doppler. Assessments are performed bilaterally. All measurements are performed with the aid of an electrocardiogram electrode.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young people;
* Young people who have followed an omnivorous diet for at least one year.

Exclusion Criteria:

* Previous alcohol or coffee abuse;
* Use of vitamin B12 supplements;
* Unstable clinical status;
* Individuals with anemia, hypertension, high cholesterol, diabetes, or a history of cardiovascular disease;
* Chronic use of medications, except oral contraceptives.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2025-05-03 (Actual)

PRIMARY OUTCOMES:
Changes in Hematological Parameters - Haemoglobin | 4 weeks
  Changes in mean hemoglobin, measured in g/dL, from baseline to 4 weeks after excluding red and processed meat from the study participants' diets.
Changes in Hematological Parameters - Reticulocytes | 4 weeks
  Changes in mean reticulocytes, measured in percentage, from baseline to 4 weeks after excluding red and processed meat from the study participants' diets.
Changes in Biochemical Parameters | 4 weeks
  Changes in mean biochemical parameters, namely Total Cholesterol, Triglycerides, HDL-C (High Density Lipoprotein Cholesterol), LDL-C (Low Density Lipoprotein Cholesterol), and Glucose, measured in mg/dL, from baseline to 4 weeks after the exclusion of red and processed meat from the study participants' diets.
Changes in Vascular Parameters - Common Carotid Artery diameters | 4 weeks
  Changes in mean systolic and mean diastolic diameters of the common carotid artery, measured in millimeters, from baseline to 4 weeks after the exclusion of red and processed meat from the diet of study participants.
Changes in Vascular Parameters - Common Carotid Artery Velocity | 4 weeks
  Changes in mean Peak Systolic velocity and Endodiastolic velocity of the common carotid artery, measured in cm/s, from baseline to 4 weeks after the exclusion of red and processed meat from the diet of study participants.
Changes in Vascular Parameters - Intima-Media Tickness | 4 weeks
  Changes in mean Intima-Media Tickness, measure in millimeters, from baseline to 4 weeks after the exclusion of red and processed meat from the diet of study participants.
Changes in Vascular Parameters - Beta Stiffness index | 4 weeks
  Changes in mean common carotid artery beta stiffness index from baseline to 4 weeks after excluding red and processed meat from the study participants' diets.
Changes in Vascular Parameters - Compliance | 4 weeks
  Changes in mean compliance, measure in mm^2. mm Hg^( -1), from baseline to 4 weeks after excluding red and processed meat from the study participants' diets.
Changes in Vascular Parameters - Heart Rate | 4 weeks
  Changes in mean heart rate, measure in bpm, from baseline to 4 weeks after excluding red and processed meat from the study participants' diets.

CONTACTS AND LOCATIONS:
Overall Officials: Helder Santos, Principal Investigator — Health School-Polytechnic Institute of Coimbra
Locations (1):
- Health School-Polytechnic Institute of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol
Time Frame: Data will be shared via the author's email.